CLINICAL TRIAL: NCT06096298
Title: Bioavailability of Vitamin B12 in Bread Using Fermented Faba Bean as B12 Source in Healthy Volunteers (BeanBread)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Anne-Maria Pajari, Associate Professor, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: BeanBread-HY
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Vitamin B12 Absorption
Keywords: cobalamin; holotranscobalamin; vitamin B12; absorption; propionibacterium freudenreichii; fermented faba bean

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study is double-masked - neither the researchers or the participants know which bread they are eating.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin B12 bread (Active Comparator): Daily dose of bread containing B12 (15 µg of vitamin B12/d) and placebo tablet (0 µg of vitamin B12/d) for 2 consecutive days.
  Interventions: Other: Vitamin B12 bread
- Positive control (Active Comparator): Daily dose of control bread (0 µg of vitamin B12/d and B12 tablet (15 µg of vitamin B12/d) for 2 consecutive days.
  Interventions: Other: Control bread
- Negative control (Placebo Comparator): Daily dose of control bread (0 µg of vitamin B12/d and placebo tablet (0 µg of vitamin B12/d) for 2 consecutive days.
  Interventions: Other: Control bread

INTERVENTIONS:
Other: Vitamin B12 bread — Wheat bread with 30 % of wheat flour replaced with fermented faba bean flour containing vitamin B12 produced by P. freudenreichii bacteria.
  Arms: Vitamin B12 bread
Other: Control bread — Wheat bread with 30 % of wheat flour replaced with fermented faba bean flour.
  Arms: Negative control; Positive control

SUMMARY:
Vitamin B12 is naturally present in animal products, but it could be added to plant-based products through fermentation using the Propionibacterium freudenreichii bacterium. This study aims to investigate the absorption of vitamin B12 synthesized by Propionibacterium freudenreichii from products made with fermented faba bean. The study products are wheat breads of which 30 % of the dry weight has been replaced with fermented faba bean flour. One of the study breads contains vitamin B12 produced by P. freudenreichii bacteria, and the other bread (control bread) is fermented using L. brevis bacteria (does not produce vitamin B12). The participants will eat the study bread for two consecutive days during the study weeks, with a washout period of 12 days. Fasting blood samples are collected on day 1 before administration of the first dose of vitamin B12 and on day 3. Nutrient intake and food consumption will be analyzed from 3-day food records at the baseline and on the bread eating days. The study is carried out in a double-blinded crossover setting.

DETAILED DESCRIPTION:
A human intervention study with healthy volunteers will be carried out to investigate the absorption of vitamin B12 synthesized by Propionibacterium freudenreichii from bread made with fermented faba bean. The study is conducted on healthy, 18-50-year-old volunteers. The study is carried out in a randomized, double-blinded, placebo-controlled crossover design.

The study products are wheat breads of which 30% of the dry weight has been replaced with fermented faba bean flour. One of the study breads contains fermented faba bean flour containing vitamin B12 produced by P. freudenreichii bacteria, and the other bread (control bread) contains faba bean flour fermented with L. brevis bacteria (does not produce vitamin B12). In addition to the study breads, the study participants are given a vitamin supplement containing cyanocobalamin as a positive control during one study week and a placebo supplement as a negative control for two weeks. During each study period, the subjects eat study breads and supplements for two consecutive days, three times a day. The study participants are otherwise allowed to follow their usual diet. On the morning of the first and third study day of each study period, a blood sample is taken from the subjects, from which the vitamin B12 bound to holotranscobalamin II and the total vitamin B12 concentration in the serum are determined. At the baseline of the study, the blood samples are also analyzed for folate, methylmalonate, homocysteine and creatinine concentrations.

Nutrient intake and food consumption will be analyzed from 3-day food records during the run-in week and each study week (total 9 days). The participants will report their gastrointestinal symptoms during the study periods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Body mass index between 18.5 and 35 kg/m2
* No exclusion criteria listed below

Exclusion Criteria:

* Food allergies against ingredients in foods supplemented in the study
* pregnancy and/or breastfeeding
* Regular use of food supplements containg B12
* Blood donation within 3 months
* Alcohol consumption more than 24 measures per week
* Smoking, using snuff
* Iron, B12 or folate deficiency
* Anemia
* small intestinal bacterial overgrowth (SIBO)
* Gastritis
* Helicobacter pylori infection
* Acid reflux
* Chron's disease
* Celiac disease
* Pancreatitis
* Abdominal surgery
* Eating disorder
* Use of supplements containing vitamin B12 in the last year
* Vitamin B12 injection treatment in the last year
* Use of metformin, protein pump inhibitors or H2-receptor blockers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12-22 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Vitamin B12 bound to transcobalamin II (holoTc) | 2 days
  Changes in serum holotranscobalamin concentrations after intake of vitamin B12
Total B12 | 2 days
  Changes in serum total B12 concentrations after intake of vitamin B12

SECONDARY OUTCOMES:
The intensity of gastrointestinal symptoms measured by a visual analogue scale | 4 weeks
  Study participants report the intensity of experienced stomach pain, cramps, bloating, flatulence, stomach noise, nausea, heartburn, unpleasant feeling and sudden need to defecate on a scale of zero (no pain at all) to 100 (very intense pain)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Maria Pajari, PhD, Principal Investigator — University of Helsinki

IPD SHARING:
Plan to Share IPD: No
The data collected is confidential and cannot be shared.